CLINICAL TRIAL: NCT07129408
Title: Epidemiological Study of the Prevalence of Mental Disorders in the Population of the Slovak Republic
Brief Title: Epidemiological Study on the Prevalence of Mental Disorders in Slovakia
Acronym: EpiMentDisSK
Status: Active, not recruiting | Type: Observational
Sponsor: Comenius University (Other)
Collaborators: European Union (Other); European Commission (Other)
Responsible Party: Principal Investigator, Alexandra Brazinova, Chair of Institute of Epidemiology, Faculty of Medicine, Comenius University
Other Study IDs: Z091007-2023
Record Dates: First submitted 2025-08-04; First posted 2025-08-19 (Actual); Last update posted 2025-08-19 (Actual); Status verified 2025-08

CONDITIONS: Depression Disorders; Bipolar Affective Disorder; Generalized Anxiety Disorder (GAD); Panic Disorder; Agoraphobia; Social Phobia; Obsessive Compulsive Disorder (OCD); Posttraumatic Stress Disorder (PTSD); Alcohol Addiction; Anorexia Nervosa; Bulimia Nervosa
Keywords: Mental disorder prevalence; Slovak Republic; Mental Health; Population study
MeSH Terms: conditions — Bipolar Disorder; Generalized Anxiety Disorder; Panic Disorder; Agoraphobia; Phobia, Social; Obsessive-Compulsive Disorder; Stress Disorders, Post-Traumatic; Alcoholism; Anorexia Nervosa; Bulimia Nervosa; Psychological Well-Being

STUDY DESIGN:
Observational Model: Other | Time Perspective: Cross-Sectional
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

SUMMARY:
This study maps the current epidemiological situation of mental disorders in Slovakia. The aim of the study is to determine the prevalence of selected mental disorders in the adult population of the Slovak Republic, assess the availability and use of mental health care services, evaluate the impact of symptoms of selected mental disorders on quality of life and functional capacity, and identify population groups at the highest risk of not using available services despite the presence of mental disorders.

The proposed project will provide unique data that have not yet been available in Slovakia on the prevalence of the most common mental disorders in the adult population in relation to age, gender, level of education, and broader social and economic contexts. It will also offer insights into the relationship between risk factors and the onset and course of these mental disorders, their overall societal impact, and the use or absence of mental health care services.

DETAILED DESCRIPTION:
Examining the current prevalence of mental disorders in the Slovak population will allow for the accurate identification of population groups who, despite experiencing symptoms of mental disorders, do not utilize mental health care services. As a result, these individuals often experience reduced functionality and a diminished quality of life. According to expert estimates, this group may include 60-80% of people with symptoms of mental disorders. However, only a population-based study that comprehensively maps this issue can provide a clear and accurate picture of the situation.

This survey on the prevalence of mental disorders and their associated risk factors will be conducted as a cross-sectional study using the internationally recognized and standardized Mini International Neuropsychiatric Interview (MINI).

The MINI instrument will be administered first to 100 respondents in a pilot phase and then to a representative sample of 3,000 respondents. Participants will be selected using a multistage sampling method that covers the entire adult population of the Slovak Republic. The selection process and data collection will be conducted by a professional research agency.

The sample size has been carefully calculated to ensure that the results are generalizable to the entire adult population of Slovakia, with a 95% confidence interval and a 2% margin of error. This representative sample will make it possible to gather sufficient data even on the least common mental disorders (with a prevalence of around 1%), ensuring that the findings are both meaningful and statistically robust.

Data collection will take place through face-to-face interviews conducted by trained interviewers from the research agency, all of whom will receive specialized training in administering the MINI tool. The data will then be subject to in-depth analysis and interpretation by experts in epidemiology, clinical psychology, sociology, and psychiatry. This multidisciplinary evaluation will serve as the foundation for developing recommendations for key ministries - including those responsible for health, education, family, and social affairs - as well as for other sectors of society. The results will also be internationally comparable, as they will align with data collected using the same methodology in other countries.

The analysis of the collected data will help identify unmet needs in mental health care, support improvements in the care of individuals with mental disorders, guide the development of a comprehensive care network, highlight at-risk population groups, and inform targeted prevention strategies.

Ultimately, this study will generate unique data - previously unavailable in Slovakia - on the prevalence of the most common mental disorders in the adult population, with regard to age, gender, educational level, and broader social and economic factors. It will also provide valuable insights into the relationship between risk factors and the development and course of mental disorders, their overall impact on society, and the accessibility and utilisation of mental health care services.

ELIGIBILITY:
Inclusion Criteria:

* age 18 years or older
* ability and willingness to undergo a face-to-face interview with an interviewer, to answer interviewer's questions from a questionnaire
* signing an informed consent

Exclusion Criteria:

* less tan 18 years

Min Age: 18 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Adult, Older Adult
Study Population: Adult population of Slovak Republic
Sampling Method: Probability Sample
Enrollment: 3100 (Actual)
Dates: Start 2025-02-13 (Actual); Primary Completion 2025-06-27 (Actual); Study Completion 2025-10-31 (Estimated)

PRIMARY OUTCOMES:
Prevalence of selected mental disorders in the Slovak Republic assessed by the Mini-International Neuropsychiatric Interview | From the end of enrolment within 6 months
  The current and lifetime prevalence of mental disorders in the Slovak population will be determined based on respondents' answers using the standardised and internationally recognised questionnaire tool, the Mini-International Neuropsychiatric Interview (MINI). Lifetime and current population prevalence and treated prevalence will be determined by age, sex, educational attainment, overall health status, social and economic determinants.

CONTACTS AND LOCATIONS:
Overall Officials: Alexandra Brazinova, prof. MD PhD, Principal Investigator — Comenius University, Faculty of Medicine, Institute of Epidemiology; Michal Hajduk, assoc.prof. PhD, Study Chair — Comenius University, Faculty of Arts, Department of Psychology; Maria Kralova, assoc.prof. MD PhD, Study Chair — Comenius University, Faculty of Medicine, Department of Psychiatry; Marek Majdan, prof. MS PhD, Study Chair — Trnava University, Faculty of Health Care and Social Work
Locations (1):
- Ministry of Health of the Slovak Republic, Bratislava, Slovakia

IPD SHARING:
Plan to Share IPD: No

REFERENCES:
- See also: Website of Ministry of Health of the Slovak Republic, informing about the study in Slovak language — https://www.health.gov.sk/Clanok?mz-studia-dusevne-poruchy